CLINICAL TRIAL: NCT03676764
Title: Community Health Azithromycin Trial in Burkina Faso
Acronym: CHAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPP1187628-A
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Childhood Mortality
Keywords: Childhood mortality; Azithromycin; Mass treatment; Vaccine Visit targeted treatment
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: All eligible communities in Nouna District will be randomized in a 1:1 fashion to biannual azithromycin or placebo. Targeted treatment (vaccine visit) will be randomized 1:1 individually to azithromycin or placebo. Randomization will be conducted by T. Porco. Procedural and algorithmic details are provided in an appendix to the Statistical Analysis Plan.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial sites will be masked to outcomes, so the responsibility for monitoring interim analysis will fall on the DSMC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Biannual mass oral azithromycin (Active Comparator): Bi-annual Mass Azithromycin distribution to all children 1-60 months old in participating communities
  Interventions: Drug: Azithromycin
- Biannual mass oral placebo (Placebo Comparator): Bi-annual Mass Placebo distribution to all children 1-60 months old in participating communities
  Interventions: Drug: Azithromycin; Drug: Placebos
- Targeted oral placebo (Placebo Comparator): Targeted placebo to children 5 to 12 weeks old at vaccine visit or other healthy child visit
  Interventions: Drug: Placebos
- Targeted oral azithromycin (Active Comparator): Targeted azithromycin to children 5 to 12 weeks old at vaccine visit or other healthy child visit
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — biannual azithromycin in eligible communities to children 1 to 59 months old Targeted azithromycin to children aged 5 to 8 weeks old at the vaccine visit
  Arms: Biannual mass oral azithromycin; Biannual mass oral placebo; Targeted oral azithromycin
Drug: Placebos — biannual placebo in eligible communities to children 1 to 59 months old Targeted placebo to children aged 5 to 8 weeks old at the vaccine visit
  Arms: Biannual mass oral placebo; Targeted oral placebo

SUMMARY:
An estimated 7.7 million pre-school aged children die each year, the majority from infectious diseases. Mass azithromycin distributions for trachoma may have the unintended benefit of reducing childhood mortality. We recently demonstrated the biannual mass azithromycin distribution significantly reduces all-cause child mortality in a cluster randomized trial (MORDOR I) conducted in three diverse regions of Sub-Saharan Africa.

Our long-term goal is to more precisely define the role of mass azithromycin treatments as an intervention for reducing childhood morbidity and mortality. We propose a cluster randomized trial designed to repeat the original study to confirm the original results in a different geographic study with similarly high child mortality, and to better understand the mechanism behind any effect of azithromycin on child mortality. We hypothesize that biannual mass azithromycin distribution will reduce child mortality compared to placebo, and that this effect will be primarily driven by a reduction in infectious burden.

Objectives:

1. Determine the efficacy of biannual mass azithromycin distribution versus placebo in children aged 1-59 months for reduction in all-cause mortality.
2. Determine the efficacy of targeted azithromycin distribution to infants during an early infant healthcare visit (approximately 5th through 12th week of life) on infant mortality.
3. Determine the mechanism behind the effect of biannual mass azithromycin distribution for reduction in child mortality.

The study will be conducted in the Nouna District in northwestern Burkina Faso.

DETAILED DESCRIPTION:
Although child health and mortality are improving worldwide, children in the Sahel and sub-Sahel regions of West Africa have the greatest risks of mortality.Burkina Faso's current under-5 mortality rate is estimated 110 per 1,000 live births. Similar to other countries in the region, the major causes of child mortality in Burkina Faso are malaria, respiratory tract infection, and diarrhea. Malnutrition acts as a major underlying contributor to mortality. Interventions that address these underlying causes may be particularly efficacious for reducing mortality.

Younger children at are at a higher risk of mortality. Approximately 2/3rd of under-5 deaths occur during the first year of life. In general, the child mortality rate decreases as age increases. While some improvement has been observed, neonatal mortality is declining at a slower rate than post-neonatal childhood mortality. Many child health interventions are designed specifically for children over 6 months of age, such as vitamin A supplementation, seasonal malaria chemoprevention, and lipid-based nutritional supplementation. Identification of strategies that are safe and effective for the youngest children will be required to address persistently high rates of neonatal and infant mortality.

The MORDOR I study demonstrated a significant reduction in all-cause child mortality following biannual mass azithromycin distribution. Across three diverse geographic locations in sub-Saharan Africa (Malawi, Niger, and Tanzania), biannual mass azithromycin distribution over a two-year period led to a 14% decrease in all-cause child mortality. In Niger, 1 in 5-6 deaths were averted. These results are qualitatively similar to those of a previous study of mass azithromycin distribution for trachoma control in Ethiopia, which found reduced odds of all-cause mortality in children in communities receiving mass azithromycin compared to control communities.

In MORDOR I, the strongest effect of azithromycin was in the youngest cohort of children. Across all three countries, the strongest effect of azithromycin was consistently in children 1-5 months of age, with an approximately 25% reduction in all-cause mortality. However, MORDOR I was not optimized to target the youngest age groups. Although children as young as 1 month were eligible, biannual distributions might not reach some children until 7 months of age. On average, children were first treated at 4 months. Given that there may be a substantial benefit to treating children at younger ages, azithromycin strategies that are designed to target younger age groups may be even more beneficial for reducing child mortality.

Here, we propose a randomized controlled trial designed to evaluate the efficacy of mass and targeted azithromycin strategies for child mortality. In the rural northwestern district of Nouna in Burkina Faso, we propose to randomize villages to biannual mass azithromycin distribution or placebo. This study was designed by CRSN and UCSF partners to confirm the results of MORDOR I, evaluate an alternative health systems distribution point (the vaccine visit) for delivery of azithromycin to young children, and to provide a platform for evaluation of potential mechanisms behind the effect of azithromycin by collecting and processing additional specimens and tests.

Objectives:

1. Determine the efficacy of biannual mass azithromycin distribution versus placebo in children aged 1-59 months for reduction in all-cause mortality.
2. Determine the efficacy of targeted azithromycin distribution to infants during an early infant healthcare visit (approximately 5th through 12th week of life) on infant mortality.
3. Determine the mechanism behind the effect of biannual mass azithromycin distribution for reduction in child mortality.

Study Design:

CRSN and UCSF (hereafter, "we") will assess childhood mortality over three years, comparing communities where children aged 1-59 months receive biannual oral azithromycin and/or targeted azithromycin during the 5th-12th week of life in conjunction with the first Expanded Programme on Immunization (EPI) vaccine visit or biannual placebo and targeted placebo. All eligible communities in Nouna District will be randomized (278 communities). A random sample of 48 (12/arm) communities from within the HDSS will be selected to participate in the "Mortality Plus" study, which will entail an annual morbidity exam among 15 randomly selected children per community to monitor infectious disease morbidity, nutritional status, and macrolide resistance. All communities will contribute to the mortality outcome.

ELIGIBILITY:
Communities:

Inclusion Criteria:

* The community location in target district.
* The community leader consents to participation in the trial (this does not obviate the need for individual consent, but without overall leadership consent, the community as a whole cannot be part of the trial).
* Eligible communities estimated population of between 200-2,000 people
* The community is not in an urban area

Exclusion criteria:

- Refusal of village chief

Individuals:

Inclusion Criteria

* All children in the study communities aged 5 to 12 weeks old at the time of the vaccination visit are eligible to participate
* Ability to feed orally
* Appropriate consent from at least one caregiver
* Family intends to stay within the study area

Exclusion Criteria:

* Individuals allergic to macrolides or azalides will not be given the study antibiotic azithromycin, but will be included in the outcome
* Refusal of parent or guardian
* Child unable to orally feed
* Family planning to move
* Children younger than 28 days old or older than 12 weeks
* Children in the bi annual drug administration group who weight less than 3.8kg.

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77664 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Oldenburg, PhD, Principal Investigator — University of California, San Francisco; Tom M Lietman, MD, Principal Investigator — University of California, San Francisco; Ali Sie, MD, PhD, Principal Investigator — Centre de Recherche en Sante de Nouna, Burkina Faso
Locations (1):
- Centre de Recherche en Sante de Nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available as per the Bill and Melinda Gates open access policy. Community based data will be available that underline the reported results (texts, tables, figures, and appendices). The study protocol and statistical analysis plan will also be made available. The data will be available following publication in accordance with the BMGF guidelines
Supporting Information: Study Protocol, SAP
Time Frame: december 2023

REFERENCES:
- [Derived] Gebreegziabher EA, Sie A, Ouattara M, Bountogo M, Coulibaly B, Boudo V, Ouedraogo T, Lebas E, Hu H, Ante-Testard PA, Gregorich SE, O'Brien KS, Hsiang MS, Glidden DV, Arnold BF, Lietman TM, Oldenburg CE. Exploring heterogeneity in treatment effects: The impact and interaction of asset-based wealth and mass azithromycin distribution on child mortality. PLoS One. 2026 Feb 9;21(2):e0341665. doi: 10.1371/journal.pone.0341665. eCollection 2026. PMID 41662252
- [Derived] Oldenburg CE, Coulibaly B, Sie A, Ouattara M, Bountogo M, Compaore G, Kiemde D, Compaore A, Zonou G, Hinterwirth A, Zhong L, Chen C, Liu Y, Yu D, Abraham T, Lebas E, Hu H, Hilde-Jones M, Arnold BF, Doan T, Lietman TM. Macrolide and non-macrolide resistance after 36 months of mass azithromycin distribution in Burkina Faso: A cluster randomized trial. Clin Infect Dis. 2026 Jan 31:ciag051. doi: 10.1093/cid/ciag051. Online ahead of print. PMID 41626759
- [Derived] Bountogo M, Ouattara M, Dah C, Coulibaly B, Ouedraogo T, Zakane A, Boudo V, Lebas E, Hu H, Arnold BF, Lietman TM, Sie A, Oldenburg CE. Azithromycin for infants at risk of poor growth and development: A pooled secondary analysis of two randomized controlled trials. PLoS One. 2025 Aug 8;20(8):e0328208. doi: 10.1371/journal.pone.0328208. eCollection 2025. PMID 40779591
- [Derived] Gebreegziabher EA, Sie A, Ouattara M, Bountogo M, Coulibaly B, Boudo V, Ouedraogo T, Lebas E, Hu H, Ante-Testard PA, Gregorich SE, O'Brien KS, Hsiang MS, Glidden DV, Arnold BF, Lietman TM, Oldenburg CE. Exploring Heterogeneity in Treatment Effects: The Impact and Interaction of Asset-Based Wealth and Mass Azithromycin Distribution on Child Mortality. medRxiv [Preprint]. 2025 Jul 6:2025.07.05.25329685. doi: 10.1101/2025.07.05.25329685. PMID 40630579
- [Derived] Gebreegziabher EA, Ouattara M, Bountogo M, Coulibaly B, Boudo V, Ouedraogo T, Lebas E, Hu H, O'Brien KS, Hsiang MS, Glidden DV, Arnold BF, Lietman TM, Sie A, Oldenburg CE. The role of Seasonal Malaria Chemoprevention in the effect of Azithromycin on Child Mortality: A Secondary Analysis of the CHAT Cluster Randomized Clinical Trial. medRxiv [Preprint]. 2025 May 2:2025.04.30.25326740. doi: 10.1101/2025.04.30.25326740. PMID 40343013
- [Derived] Sie A, Ouattara M, Bountogo M, Boudo V, Ouedraogo T, Dah C, Compaore G, Lebas E, Hu H, Porco TC, Arnold BF, O'Brien KS, Lietman TM, Oldenburg CE. Mass azithromycin for prevention of child mortality among children with acute malnutrition: A subgroup analysis of a cluster randomized controlled trial. PLOS Glob Public Health. 2024 Oct 28;4(10):e0003875. doi: 10.1371/journal.pgph.0003875. eCollection 2024. PMID 39466816
- [Derived] Oldenburg CE, Ouattara M, Bountogo M, Boudo V, Ouedraogo T, Compaore G, Dah C, Zakane A, Coulibaly B, Bagagnan C, Hu H, O'Brien KS, Nyatigo F, Keenan JD, Doan T, Porco TC, Arnold BF, Lebas E, Sie A, Lietman TM. Mass Azithromycin Distribution to Prevent Child Mortality in Burkina Faso: The CHAT Randomized Clinical Trial. JAMA. 2024 Feb 13;331(6):482-490. doi: 10.1001/jama.2023.27393. PMID 38349371
- [Derived] Sie A, Ouattara M, Bountogo M, Dah C, Ouedraogo T, Boudo V, Lebas E, Hu H, Arnold BF, O'Brien KS, Lietman TM, Oldenburg CE. Single-dose azithromycin for infant growth in Burkina Faso: Prespecified secondary anthropometric outcomes from a randomized controlled trial. PLoS Med. 2024 Jan 23;21(1):e1004345. doi: 10.1371/journal.pmed.1004345. eCollection 2024 Jan. PMID 38261579
- [Derived] Sie A, Ouattara M, Bountogo M, Boudo V, Ouedraogo T, Compaore G, Dah C, Bagagnan C, Lebas E, Hu H, Rice J, Porco TC, Arnold BF, Lietman TM, Oldenburg CE. Azithromycin during Routine Well-Infant Visits to Prevent Death. N Engl J Med. 2024 Jan 18;390(3):221-229. doi: 10.1056/NEJMoa2309495. PMID 38231623
- [Derived] Sie A, Ouattara M, Bountogo M, Bagagnan C, Coulibaly B, Boudo V, Lebas E, Brogdon JM, Lin Y, Barnighausen T, Porco TC, Doan T, Lietman TM, Oldenburg CE; Etude CHAT Study Group. A double-masked placebo-controlled trial of azithromycin to prevent child mortality in Burkina Faso, West Africa: Community Health with Azithromycin Trial (CHAT) study protocol. Trials. 2019 Dec 4;20(1):675. doi: 10.1186/s13063-019-3855-9. PMID 31801563

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Cluster
Period: Overall Study
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo | Targeted Oral Azithromycin | Targeted Oral Placebo
Started (For the cluster randomization trial (first two arm), we have census at timepoint 0, 6, 12, 18, 24, 30, 36. The randomization units are cluster/community. For the individual randomization trial (last two arm), we have baseline and 6 month. The randomization units are children/participants.) | 22148; 144 Cluster (Cluster Randomized; Unit: cluster/community) | 22639; 140 Cluster (Cluster Randomized; Unit: cluster/community) | 16416; 0 Cluster (Individual Randomized; Unit: children/participant) | 16461; 0 Cluster (Individual Randomized; Unit: children/participant)
Completed (In the first two arm, number of children in last census (census at month 36) were reported.) | 19924; 132 Cluster (Cluster Randomized; Unit: cluster/community) | 19351; 126 Cluster (Cluster Randomized; Unit: cluster/community) | 15734; 0 Cluster (Individual Randomized; Unit: children/participant) | 15701; 0 Cluster (Individual Randomized; Unit: children/participant)
Not Completed | 2224; 12 Cluster | 3288; 14 Cluster | 682; 0 Cluster | 760; 0 Cluster

BASELINE CHARACTERISTICS:
Population: The units are all participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo | Targeted Oral Azithromycin | Targeted Oral Placebo | Total
Number analyzed (Participants) | 22148 | 22639 | 16416 | 16461 | 77664
Age, Continuous [Median (Standard Deviation); unit: month] | 31 (16.71) | 31 (16.71) | 1.51 (0.51) | 1.55 (0.51) | 10 (19.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10883 | 11249 | 8045 | 8136 | 38313
  Male | 11265 | 11390 | 8371 | 8325 | 39351
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 22148 | 22639 | 16416 | 16461 | 77664
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 22148 | 22639 | 16416 | 16461 | 77664

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Rate in Children Aged 1-59 Months
Description: All-cause mortality as determined by biannual census among children aged 1-59 months
Time Frame: 36 months
Population: Primary analysis included 34399 children in azithromycin clusters and 33847 children placebo clusters during 6 census periods. Person-time for the denominator was calculated by summing the person-time for each intercensal period. Children who were alive during both censuses contributed the person-time for that intercensal period. A cluster that was not censused, eg, due to security, could reenter the study at a later census.
Measure: Number; unit: deaths per 1000 person years
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 34399 | 33847
deaths per 1000 person years | 8.2 | 10.0

2. Primary Outcome: All-cause Mortality Rate in Individually Randomized Children at 4-12 Weeks of Age
Description: All-cause mortality as determined by a follow-up visit for individually randomized children at healthy child visits
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Oral Azithromycin | Targeted Oral Placebo
Number analyzed (Participants) | 15734 | 15701
Participants | 82 | 75

3. Secondary Outcome: Malaria Parasitemia in Children 1-59 Months at 36 Months
Description: Malaria parasitemia as measured by thin and thick smears in a random sample of children at 36 months
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 345 | 344
Participants | 90 | 114

4. Secondary Outcome: Weight-for-height Z-score in Individually Randomized Children at Healthy Child Visits
Description: The WHZ is calculated using weight (kg) and height (cm) measurements taken at healthy child visits and converted into Z-scores using the WHO Growth Standards. Z-scores represent the number of standard deviations from the median of a reference population.
  A WHZ of 0 represents the median of the reference population, while negative Z-scores indicate below-average weight-for-height, and positive Z-scores indicate above-average weight-for-height. A WHZ below -2 is indicative of wasting, while a WHZ above +2 is considered overweight.
Time Frame: 6 months
Population: 13641 children in Targeted oral azithromycin arm and 13657 children in Targeted oral placebo arm had valid height and weight measurement
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Targeted Oral Azithromycin | Targeted Oral Placebo
Number analyzed (Participants) | 13641 | 13567
z-score | -0.64 (1.2) | -0.64 (1.2)

5. Secondary Outcome: Height-for-age Z-score in Individually Randomized Children at Healthy Child Visits
Description: The Height-for-age Z-score (HAZ) is calculated using height (cm) measurements taken at healthy child visits and converted into Z-scores using the WHO Growth Standards. Z-scores represent the number of standard deviations from the median of a reference population.
  A HAZ of 0 represents the median of the reference population, while negative Z-scores indicate below-average height-for-age, and positive Z-scores indicate above-average height-for-age. A HAZ below -2 is indicative of stunting, reflecting chronic undernutrition or growth failure.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Targeted Oral Azithromycin | Targeted Oral Placebo
Number analyzed (Participants) | 13641 | 13657
z score | -0.31 (1.3) | -0.31 (1.3)

6. Secondary Outcome: Mid-upper Arm Circumference in Individually Randomized Children at Healthy Child Visits
Time Frame: 6 months
Population: 13641 children in azithromycin group and 13657 children in placebo group had valid MUAC measurement at 6 month
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Targeted Oral Azithromycin | Targeted Oral Placebo
Number analyzed (Participants) | 13641 | 13657
cm | 13.8 (1.2) | 13.8 (1.2)

7. Secondary Outcome: Linear Growth in Individually Randomized Children
Description: Change in length per day from baseline to 6 months
Time Frame: 6 months
Population: 13641 children in azithromycin group and 13657 children in placebo group had valid length measurement at 6 month
Measure: Mean (Standard Deviation); unit: mm/day
Arm/Group | Targeted Oral Azithromycin | Targeted Oral Placebo
Number analyzed (Participants) | 13641 | 13657
mm/day | 8.0 (2.1) | 8.0 (2.3)

8. Secondary Outcome: Weight Gain in Individually Randomized Children
Description: Change in weight per day from baseline to 6 months
Time Frame: 6 months
Population: 13641 children in azithromycin group and 13657 children in placebo group had valid weight measurement at 6 month
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Targeted Oral Azithromycin | Targeted Oral Placebo
Number analyzed (Participants) | 13641 | 13657
g/day | 18 (6.2) | 18 (6.4)

ADVERSE EVENTS:
Time Frame: For the Biannual Mass Oral Azithromycin/Placebo arm, adverse events among infants <6 months of age participating in the first treatment round in a subset of 48 study clusters. Adverse events were collected 2 weeks following the distribution of azithromycin or placebo. For Targeted Oral Azithromycin/Placebo arm, active surveillance for adverse events was performed in a random sample of 10% of enrolled infants and recorded at 2 weeks after administration of azithromycin or placebo.
Description: All-cause mortality was monitored at every census/visit in all arms. The number at risk for mortality reflects children included over the study period.
  Adverse events (AEs) were collected for 2 weeks post-distribution: in all selected clusters for Biannual Mass Az/Pl arms and a 10% random sample in the Targeted Az/Pl arm. The number at risk for AEs refers to children completing the 2-week follow-up, which differs from the Participant Flow module.
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo | Targeted Oral Azithromycin | Targeted Oral Placebo
All-Cause Mortality (participants affected / at risk) | 498/34399 | 588/33847 | 82/16416 | 75/16461
Serious Adverse Events (participants affected / at risk) | 0/269 | 0/199 | 5/1606 | 1/1532
Other Adverse Events (participants affected / at risk) | 77/269 | 14/199 | 62/1606 | 79/1532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biannual Mass Oral Azithromycin (N=269) | Biannual Mass Oral Placebo (N=199) | Targeted Oral Azithromycin (N=1606) | Targeted Oral Placebo (N=1532)
Death (General disorders) | 0 | 0 | 0 | 1
Hospitalization (General disorders) | 0 | 0 | 5 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biannual Mass Oral Azithromycin (N=269) | Biannual Mass Oral Placebo (N=199) | Targeted Oral Azithromycin (N=1606) | Targeted Oral Placebo (N=1532)
Diarrhea (Gastrointestinal disorders) | 30 | 5 | 36 | 45
Abdominal pain (General disorders) | 19 | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 0 | 24 | 38
Constipation (Gastrointestinal disorders) | 10 | 0 | 9 | 14
Hemorrhoids (Gastrointestinal disorders) | 5 | 3 | 6 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03676764/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03676764/SAP_001.pdf